CLINICAL TRIAL: NCT03321149
Title: RiseTx: Testing the Feasibility of a Web Application for Reducing Sedentary Behavior Among Prostate Cancer Survivors Receiving Androgen Deprivation Therapy
Brief Title: Reducing Sedentary Behavior Among Prostate Cancer Survivors on Androgen Deprivation Therapy
Acronym: RiseTx
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Collaborators: University of Toronto (Other); Toronto Sunnybrook Regional Cancer Centre (Other); Princess Margaret Hospital, Canada (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB2017
Record Dates: First submitted 2017-10-12; First posted 2017-10-25 (Actual); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Prostate Cancer; Prostate Neoplasm; Cancer; Sedentary Lifestyle
Keywords: Web-based intervention; Sedentary behavior; Lifestyle intervention; Feasibility
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms; Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RiseTx (Experimental): Participants were given access to the RiseTx application and an activity monitor to participate in the five phase intervention.
  Interventions: Other: RiseTx

INTERVENTIONS:
Other: RiseTx — Participants were given access to the RiseTx application, as well as given a Jawbone, a wrist-worn device that can assess activity patterns throughout the day and provide sensory alerts to stand after prolonged sitting (i.e., ≥30 minutes of sedentary time). The intervention consisted of five phases following initial data collection that comprised of self-regulatory strategies to reduce sitting time and self-monitoring of step counts.

SUMMARY:
The current study aimed to develop and assess an easy-to-use, highly accessible mobile and web-based application intervention to reduce sedentary behavior and increase physical activity in the hope of reducing the side effects of treatment and improving quality of life for the 13,000 or more prostate cancer survivors who are prescribed ADT each year in Canada. The study was conducted in two phases, where Phase one was focused on finding out about the attitudes and perceptions of sedentary behavior and the use of mobile applications among prostate cancer survivors using semi-structured interviews. Together with professional experts and a group of men who were diagnosed with prostate cancer, we developed RiseForTx - an application that is used on a smartphone or tablet to reduce time spent in, and to change patterns of, sedentary behaviour each day (Phase two). Part of the intervention was also focused on increasing daily steps to improve physical activity. We tested the intervention to examine (i) how the application works, (ii) if prostate cancer survivors like it and use it; and (iii) if sedentary behaviour and physical activity can reduce the impact of the side effects for treatment and improve quality of life among men on ADT.

DETAILED DESCRIPTION:
In the first 10 days following recruitment, participants met with the research coordinator and were provided with an accelerometer (GT3X) and completed self-report baseline measures. Provided along with the RiseTx application is the Jawbone, which is a wrist-worn device that can assess activity patterns throughout the day and provide sensory alerts to stand after prolonged sitting (i.e., ≥30 minutes of sedentary time). The intervention consisted of five phases following initial data collection, including a baseline phase (weeks 1-2) where participants self-monitored their typical leisure time PA (i.e., step counts) and were asked to 'sync' their Jawbone with the RiseTx application to view their daily progress and steps. This daily self-monitoring process continued over the remaining intervention period. Based on a previously tested ramped step count approach that focuses on increasing walking by an extra 1000 daily steps over a set period, participants attempted to increase daily steps by 1000 over the average of their baseline week. Phases I-III involved progressive release of self-regulatory strategies (e.g., action planning) on the application and targeted changes in both sitting time (and breaks in sitting time) and step counts. Phase I (weeks 3-4) focused on increasing low intensity, incidental movement, through the use of an alerting device, and the Jawbone (reminder to break SED). At this time, an additional +1000 daily step increment was set above baseline. Phase II (weeks 5-6) targeted shorter planned PA (of up to 10 mins) by having participants form action plans on the application for both reducing SED and increasing PA. An additional +1000 daily step increment was set above Phase I. Phase III (weeks 7-8) focused on promoting longer, moderate intensity PA (>10 min), where participants used the application to form coping plans for barriers to reducing sitting time or engaging in PA. An additional +1000 daily step increment was set above Phase II step target. A 4-week consolidation phase (Phase IV and V; weeks 9-12) followed, where participants received weekly reminders that encouraged them to continue to use the RiseTx application to practice combining the different self-regulatory strategies learned in Phases I-III. Following the intervention, there was a 12-week maintenance period (weeks 13-24) where participants no longer received weekly self-regulatory practice reminders, yet still had access to the application.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Men with localized or asymptomatic metastatic primary prostate cancer (Stage I-III)
* Currently receiving ADT (continuous and/or intermittent) for at least 6 months
* Active e-mail address to access the intervention website
* Proficient in English
* Physically inactive (< 150 minutes of moderate-intensity PA/week)
* No uncontrolled co-morbidities
* Medical clearance from the primary healthcare provider

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2016-10-01 (Actual); Study Completion 2016-10-01 (Actual)

PRIMARY OUTCOMES:
Feasibility measures | 12 weeks
  Intervention adherence was tracked through website analytics such as number of logins (≥ 3 visits by participants each week to the RiseTx platform)

SECONDARY OUTCOMES:
Physical Activity (PA) | Baseline, 12 Weeks, 24 week follow-up
  PA was measured by ActiGraph Model GT3X accelerometers
Step counts | Baseline and 12 Weeks
  Weekly step counts were collected using the Jawbone UP24.
Sedentary Behavior (SED) | Baseline, 12 Weeks, 24 week follow-up
  Volume of SED was measured by ActiGraph Model GT3X accelerometers.
Quality of life | Baseline, 12 Weeks, 24 week follow-up
  Quality of life was assessed by the validated Functional Assessment of Cancer Therapy-General (FACT-G).
Cancer-specific quality of life | Baseline, 12 Weeks, 24 week follow-up
  FACT-Prostate contains 12 questions that assess the most important targeted symptoms and concerns for participants.

OTHER OUTCOMES:
Feasibility measures | Baseline, 12 Weeks, 24 week follow-up
  Measurement completion was assessed by evaluating whether ≥75% of participants completed baseline, 12-weeks, and 24-week follow-up measures
Feasibility measures | 12 Weeks
  Acceptability was measured through an intervention satisfaction survey completed at post-intervention assessing perceptions and overall impressions of the RiseTx intervention (>75% rate their participation as satisfactory or very satisfactory)
Feasibility measures | Baseline, 12 Weeks, and 24 week follow-up
  Attrition was assessed by evaluating whether there was a ≤20% drop-out rate

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gilson ND, Faulkner G, Murphy MH, Meyer MR, Washington T, Ryde GC, Arbour-Nicitopoulos KP, Dillon KA. Walk@Work: An automated intervention to increase walking in university employees not achieving 10,000 daily steps. Prev Med. 2013 May;56(5):283-7. doi: 10.1016/j.ypmed.2013.01.022. Epub 2013 Feb 13. PMID 23415624
- [Background] Mitchell MS, Goodman JM, Alter DA, John LK, Oh PI, Pakosh MT, Faulkner GE. Financial incentives for exercise adherence in adults: systematic review and meta-analysis. Am J Prev Med. 2013 Nov;45(5):658-67. doi: 10.1016/j.amepre.2013.06.017. PMID 24139781
- [Background] Arain M, Campbell MJ, Cooper CL, Lancaster GA. What is a pilot or feasibility study? A review of current practice and editorial policy. BMC Med Res Methodol. 2010 Jul 16;10:67. doi: 10.1186/1471-2288-10-67. PMID 20637084
- [Background] Kuijpers W, Groen WG, Aaronson NK, van Harten WH. A systematic review of web-based interventions for patient empowerment and physical activity in chronic diseases: relevance for cancer survivors. J Med Internet Res. 2013 Feb 20;15(2):e37. doi: 10.2196/jmir.2281. PMID 23425685
- [Background] Cella DF, Tulsky DS, Gray G, Sarafian B, Linn E, Bonomi A, Silberman M, Yellen SB, Winicour P, Brannon J, et al. The Functional Assessment of Cancer Therapy scale: development and validation of the general measure. J Clin Oncol. 1993 Mar;11(3):570-9. doi: 10.1200/JCO.1993.11.3.570. PMID 8445433
- [Background] Esper P, Mo F, Chodak G, Sinner M, Cella D, Pienta KJ. Measuring quality of life in men with prostate cancer using the functional assessment of cancer therapy-prostate instrument. Urology. 1997 Dec;50(6):920-8. doi: 10.1016/S0090-4295(97)00459-7. PMID 9426724
- [Background] Leon AC, Davis LL, Kraemer HC. The role and interpretation of pilot studies in clinical research. J Psychiatr Res. 2011 May;45(5):626-9. doi: 10.1016/j.jpsychires.2010.10.008. Epub 2010 Oct 28. PMID 21035130
- [Derived] Trinh L, Arbour-Nicitopoulos KP, Sabiston CM, Berry SR, Loblaw A, Alibhai SMH, Jones JM, Faulkner GE. RiseTx: testing the feasibility of a web application for reducing sedentary behavior among prostate cancer survivors receiving androgen deprivation therapy. Int J Behav Nutr Phys Act. 2018 Jun 7;15(1):49. doi: 10.1186/s12966-018-0686-0. PMID 29880049